CLINICAL TRIAL: NCT03131505
Title: Perspectives on the INternational CLassification of Diseases (11th Revision); Using Lived Experience to Improve Mental Health Diagnosis in NHS England: INCLUDE Study
Brief Title: INCLUDE: Using Lived Experience to Improve Mental Health Diagnosis v1
Acronym: INCLUDE
Status: Completed | Type: Observational
Sponsor: Norfolk and Suffolk NHS Foundation Trust (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: 216352
Record Dates: First submitted 2017-04-20; First posted 2017-04-27 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Mental Health Issue (E.G., Depression, Psychosis, Personality Disorder, Substance Abuse); Schizophrenia; Generalised Anxiety Disorder; Bipolar Disorder
MeSH Terms: conditions — Depression; Psychotic Disorders; Personality Disorders; Substance-Related Disorders; Schizophrenia; Generalized Anxiety Disorder; Bipolar Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The focus of this study is not about what it is like to have a mental disorder, but instead the diagnostic experience.

Some people find diagnoses helpful, but some find them upsetting and harmful. Research is therefore needed to improve diagnostic processes. It has been suggested that patient experiences and outcomes may be affected by the diagnostic tools used, including diagnostic criteria, labels and language. In the NHS, the tool used by doctors to help diagnose people is a guidebook called the International Classification of Diseases (ICD). A new version of this guide is due to be released in 2018.

This project will use focus groups to ask people who use mental health services and diagnosing doctors in those services what they think about the labels and language in the new guide. The investigators can then suggest changes before the guide is published. The investigators hope that this research will improve mental health diagnosis. The research will take place in Norfolk and Suffolk and span eight months.

DETAILED DESCRIPTION:
This is a qualitative project requested by the World Health Organisation (WHO), and planned by Norfolk and Suffolk NHS Foundation Trust and the University of East Anglia. The research aims and design have been developed in consultation with service users, clinicians, academics and the World Health Organisation (WHO). These groups have told the investigators that mental health diagnosis can have unintended, negative consequences. This is supported by a large body of existing research. It has been suggested that patient experiences and outcomes may be affected by the diagnostic classifications used (i.e. labels and language). The investigators plan to explore service users' and clinicians' views on the proposed ICD-11 diagnostic classifications. To do this, the investigators will provide participants with the proposed ICD-11 diagnostic classification relevant to their experience, and conduct focus groups to explore people's views of the new diagnostic classifications, including judgement about the clinical accuracy, the language used, what people think is helpful and unhelpful, and what could be improved. The topic guide for the focus groups will be developed in consultation with the advisory group (comprising service users, carers and clinicians).

The investigators will conduct separate focus groups for service users and clinicians as the investigators believe joint groups may impact the findings. The investigators will collate findings to produce recommendations for the criteria and language proposed for ICD-11. These recommendations will be discussed in feedback groups of service users, carers and clinicians, which will provide further participants an opportunity for additional thoughts and reflection.

Inclusion

* Adult service users will have formally received one of the five diagnoses under investigation: Unipolar Depression,Schizophrenia, Bipolar Disorder, Generalised Anxiety Disorder or Personality Disorder.
* Individuals will be excluded if their participation is deemed unsafe to themselves or others by their clinical team or clinicians on the research team.
* Clinicians will have had experience working with mental health, either as a GP or psychiatrist, where diagnosing one of the above five diagnoses is part of their role.
* Carers will have had experience looking after someone diagnosed with one of the five diagnoses mentioned above.
* Participants who have been involved in one aspect of the study will be excluded from taking part in any other aspects (e.g. participants in the focus group may not be involved in other focus or feedback groups).
* Participants with multiple diagnoses will only be allowed to attend one focus group, but they may choose which one of the relevant focus groups they would like to take part in.

Exclusion:

* Non-English speakers will not be included in the study.
* Individuals under 18 years old will be excluded.
* Individuals who do not have capacity to give consent will be excluded. Individuals who lose capacity at any point between referral and the end of their participation will be removed from the study.

ELIGIBILITY:
Inclusion:

1. Adult service users will have formally received one of the five diagnoses under investigation: Unipolar Depression, Schizophrenia, Bipolar Disorder, Generalised Anxiety Disorder or Personality Disorder.
2. Clinicians will have had experience working with mental health, either as a GP or psychiatrist, where diagnosing any of the above diagnoses is part of their role.
3. Carers will have had experience looking after someone with the above diagnoses.
4. Service users with multiple diagnoses will be allowed to participate, and choose which one of the relevant focus groups they would like to attend.
5. Service users will be under the care of an NSFT service.

Exclusion:

1. Individuals under 18 years old.
2. Individuals who do not have capacity to give consent.
3. Individuals who lose capacity during the study.
4. Individuals who do not speak English.
5. Individuals will be excluded if their participation is deemed unsafe to themselves or others by their lead clinician or clinicians on the research team.
6. Individuals who have taken part in another group or part of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mental health service users clinicians
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Qualitative evaluation of the impact of new ICD-11 diagnostic criteria via focus groups with people living with mental health conditions and clinicians. | 8 months
  Focus groups will be undertaken with people who have received a mental health diagnosis (unipolar or bipolar depression, generalised anxiety disorder, schizophrenia, personality disorder) and clinicians working in mental health services. The focus groups will follow a structured topic guide, based around the new diagnostic criteria and language for each condition to understand participants' views on meaning, accessibility, stigma and recovery

CONTACTS AND LOCATIONS:
Overall Officials: Corinna Hackmann, Principal Investigator — Norfolk and Suffolk NHS Foundation Trust
Locations (1):
- Norfolk and Suffolk NHS Foundation Trust, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hackmann C, Green A, Notley C, Perkins A, Reed GM, Ridler J, Wilson J, Shakespeare T. Protocol for a qualitative study exploring perspectives on the INternational CLassification of Diseases (11th revision); Using lived experience to improve mental health Diagnosis in NHS England: INCLUDE study. BMJ Open. 2017 Sep 3;7(9):e018399. doi: 10.1136/bmjopen-2017-018399. PMID 28871029